CLINICAL TRIAL: NCT01987960
Title: Interventional, Randomised, Double-blind, Parallel-group, Placebo-controlled, Flexible-dose Study of Brexpiprazole as Adjunctive Treatment to Paroxetine or Sertraline in Adult Patients Suffering From Post-traumatic Stress Disorder (PTSD)
Brief Title: Brexpiprazole as an Adjunctive Treatment to Paroxetine or Sertraline in Adult Patients Suffering From Post-traumatic Stress Disorder (PTSD)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated due to challenges with patient eligibility; the decision to terminate was not based on any safety concerns
Sponsor: H. Lundbeck A/S (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14865A; 2012-004982-41 (EudraCT Number)
Record Dates: First submitted 2013-11-13; First posted 2013-11-20 (Estimated); Results first posted 2017-03-13 (Actual); Last update posted 2017-03-13 (Actual); Status verified 2017-01

CONDITIONS: Post-traumatic Stress Disorder; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — brexpiprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo adjunct to open-label treatment with a commercially available approved treatment for PTSD (PAR/SER)
  Interventions: Drug: Placebo
- Brexpiprazole (Experimental): Brexpiprazole adjunct to open-label treatment with a commercially available approved treatment for PTSD (PAR/SER). Brexpiprazole dosing was 1mg/day for one week, followed by 2mg/day for 3 weeks. Thereafter the dose was flexible and could be adjusted from 1 to 3 mg/day.
  Interventions: Drug: Brexpiprazole

INTERVENTIONS:
Drug: Placebo — Once daily, tablets, orally
  Arms: Placebo
Drug: Brexpiprazole — 1 to 3 mg/day, once daily dose, tablets, orally
  Arms: Brexpiprazole

SUMMARY:
To evaluate the efficacy of brexpiprazole as adjunctive treatment to paroxetine (PAR) or sertraline (SER) on PTSD symptoms.

ELIGIBILITY:
Inclusion Criteria:

* The patient has PTSD, diagnosed according to DSM-IV-TR™ and confirmed by the Mini International Neuropsychiatric Interview (MINI).
* The patient has a Clinician-Administered PTSD Scale Part 2 (CAPS-2) total score ≥70 at Screening and Baseline Visits.
* The reported duration of the PTSD is at least 3 months.

Exclusion Criteria:

* The index traumatic event that led to development of PTSD took place more than 15 years before screening.
* The patient has a severe personality disorder that in the investigator's opinion may interfere with the conduct of the study.
* The patient is at significant suicidal risk.

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 417 (Actual)
Dates: Start 2013-12; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (59):
- United States (22):
  - US004, Los Angeles, California
  - US025, Los Angeles, California
  - US024, Riverside, California
  - US015, San Diego, California
  - US008, San Diego, California
  - US002, Bradenton, Florida
  - US006, Gainesville, Florida
  - US016, Jacksonville, Florida
  - US020, North Miami, Florida
  - US017, Tampa, Florida
  - US012, Indianapolis, Indiana
  - US021, Roslindale, Massachusetts
  - US019, Las Vegas, Nevada
  - US007, Nashua, New Hampshire
  - US001, The Bronx, New York
  - US009, Cincinnati, Ohio
  - US005, Dayton, Ohio
  - US010, Portland, Oregon
  - US014, Norristown, Pennsylvania
  - US011, Memphis, Tennessee
  - US003, Austin, Texas
  - US026, Seattle, Washington
- EE001, Tallinn, Estonia
- Finland (6):
  - FI002, Helsinki
  - FI003, Helsinki
  - FI001, Kuopio
  - FI006, Oulu
  - FI005, Tampere
  - FI004, Turku
- France (5):
  - FR002, Fort de France
  - FR003, Laxou
  - FR004, Nîmes
  - FR005, Thuir
  - FR001, Tours
- Italy (5):
  - IT005, Andria
  - IT004, Catania
  - IT003, Lecce
  - IT001, Pisa
  - IT002, Siena
- Poland (5):
  - PL003, Bialystok
  - PL004, Gdansk
  - PL005, Gdansk
  - PL001, Leszno
  - PL002, Lublin
- Serbia (3):
  - RS006, Belgrade
  - RS004, Niš
  - RS005, Novi Kneževac
- South Africa (9):
  - ZA006, Bloemfontein
  - ZA002, Cape Town
  - ZA003, Cape Town
  - ZA004, Cape Town
  - ZA005, Cape Town
  - ZA008, Durban
  - ZA007, Port Elizabeth
  - ZA001, Pretoria
  - ZA009, Pretoria
- Sweden (3):
  - SE001, Falun
  - SE002, Stockholm
  - SE003, Uppsala

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 417 patients were enrolled to the study and 413 patients received open-label treatment with a commercially available treatment for PTSD (PAR/SER) in Period 1. Only 40 patients were randomized to Period 2, the randomized period, before the study was terminated; 190 patients entered Period 3. Data are only reported for the randomized period.
Groups:
- Period 1 Placebo and PAR/SER: Placebo adjunct to open-label treatment with a commercially available approved treatment for PTSD (PAR/SER).
  Placebo: Once daily, tablets, orally
- Period 2 Placebo and PAR/SER (Randomized Period): Randomized placebo adjunct to open-label treatment with a commercially available approved treatment for PTSD (PAR/SER); randomized period.
  Placebo: Once daily, tablets, orally
- Period 2 Brexpiprazole and PAR/SER (Randomized Period): Randomized brexpiprazole adjunct to open-label treatment with a commercially available approved treatment for PTSD (PAR/SER). Brexpiprazole dosing was 1mg/day for one week, followed by 2mg/day for 3 weeks. Thereafter the dose was flexible and could be adjusted from 1 to 3 mg/day; randomized period
  Brexpiprazole: 1 to 3 mg/day, once daily dose, tablets, orally
- Period 3 Placebo and PAR/SER: Continuation of treatment with placebo adjunct to open-label treatment with a commercially available approved treatment for PTSD (PAR/SER) from Period 1.
  Placebo: Once daily, tablets, orally
Period: Period 1
Arm/Group | Period 1 Placebo and PAR/SER | Period 2 Placebo and PAR/SER (Randomized Period) | Period 2 Brexpiprazole and PAR/SER (Randomized Period) | Period 3 Placebo and PAR/SER
Started | 417 | 0 | 0 | 0
Completed | 231 | 0 | 0 | 0
Not Completed | 186 | 0 | 0 | 0
Not completed — Adverse Event | 24 | 0 | 0 | 0
Not completed — Lack of Efficacy | 4 | 0 | 0 | 0
Not completed — Non-compliance with IMP | 6 | 0 | 0 | 0
Not completed — Protocol Violation | 12 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 21 | 0 | 0 | 0
Not completed — Lost to Follow-up | 40 | 0 | 0 | 0
Not completed — administrative or other reason | 75 | 0 | 0 | 0
Not completed — Withdrawal of consent before treatment | 4 | 0 | 0 | 0
Period: Period 2
Arm/Group | Period 1 Placebo and PAR/SER | Period 2 Placebo and PAR/SER (Randomized Period) | Period 2 Brexpiprazole and PAR/SER (Randomized Period) | Period 3 Placebo and PAR/SER
Started | 0 | 17 | 23 | 0
Completed | 0 | 12 | 14 | 0
Not Completed | 0 | 5 | 9 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Administrative or other reason | 0 | 5 | 7 | 0
Period: Period 3
Arm/Group | Period 1 Placebo and PAR/SER | Period 2 Placebo and PAR/SER (Randomized Period) | Period 2 Brexpiprazole and PAR/SER (Randomized Period) | Period 3 Placebo and PAR/SER
Started | 0 | 0 | 0 | 190
Completed | 0 | 0 | 0 | 119
Not Completed | 0 | 0 | 0 | 71
Not completed — Adverse Event | 0 | 0 | 0 | 7
Not completed — Non-compliance with IMP | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 9
Not completed — Lost to Follow-up | 0 | 0 | 0 | 5
Not completed — Administrative or other reason | 0 | 0 | 0 | 43

BASELINE CHARACTERISTICS:
Population: The all-patients-treated set (APTS) comprises all randomized patients who took at least one dose of brexpiprazole or placebo.
Groups:
- Period 2 Brexpiprazole and PAR/SER (Randomized Period): Randomized brexpiprazole adjunct to open-label treatment with a commercially available approved treatment for PTSD (PAR/SER). Brexpiprazole dosing was 1mg/day for one week, followed by 2mg/day for 3 weeks. Thereafter the dose was flexible and could be adjusted from 1 to 3 mg/day; randomized period.
  Brexpiprazole: 1 to 3 mg/day, once daily dose, tablets, orally
- Total: Total of all reporting groups
Arm/Group | Period 2 Placebo and PAR/SER (Randomized Period) | Period 2 Brexpiprazole and PAR/SER (Randomized Period) | Total
Number analyzed (Participants) | 17 | 23 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (11.8) | 47.6 (10.4) | 45.6 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 7 | 12 | 19

OUTCOME MEASURES:

1. Primary Outcome: PTSD Symptoms Using CAPS-2 Total Score
Description: Clinician-Administered PTSD Scale Part 2 (CAPS-2): 17 items in criteria B, C and D (Corresponding to CAPS-2) will be administered to provide a total score. They are rated on a 5 point scale for frequency from 0 (never or none) to 4 (daily or almost every day), and intensity from 0 (none) to 4 (extreme). The sum of the 17 items gives a toal score ranging from 0 to 136, with a higher score indicating greater symptom severity.
Time Frame: Period 2: Baseline to Week 12 (of randomized period)
Population: Due to the low number of enrolled patients eligible for randomization and the sponsor's early termination of the study, the data presented are descriptive i.e. the primary and key secondary efficacy analyses were not done
Measure: Mean (Standard Deviation); unit: Score
Groups:
- Period 2 Absolute Mean at Baseline; Placebo and PAR/SER: Period 2 absolute mean value at Baseline; Randomized placebo adjunct to open-label treatment with a commercially available approved treatment for PTSD (PAR/SER); randomized period.
  Placebo: Once daily, tablets, orally
- Period 2 Absolute Mean at Baseline; Brexpiprazole and PAR/SER: Period 2 absolute mean value at Baseline; Randomized brexpiprazole adjunct to open-label treatment with a commercially available approved treatment for PTSD (PAR/SER). Brexpiprazole dosing was 1mg/day for one week, followed by 2mg/day for 3 weeks. Thereafter the dose was flexible and could be adjusted from 1 to 3 mg/day; randomized period.
  Brexpiprazole: 1 to 3 mg/day, once daily dose, tablets, orally
- Period 2 Absolute Mean at Week 12; Placebo and PAR/SER: Period 2 absolute mean value at Week 12; Randomized placebo adjunct to open-label treatment with a commercially available approved treatment for PTSD (PAR/SER); randomized period.
  Placebo: Once daily, tablets, orally
  Absolute values at Week 12 in Period 2 (Study Week 24)
- Period 2 Absolute Mean at Week 12; Brexpiprazole and PAR/SER: Period 2 absolute mean value at Week 12; Randomized brexpiprazole adjunct to open-label treatment with a commercially available approved treatment for PTSD (PAR/SER). Brexpiprazole dosing was 1mg/day for one week, followed by 2mg/day for 3 weeks. Thereafter the dose was flexible and could be adjusted from 1 to 3 mg/day; randomized period.
  Brexpiprazole: 1 to 3 mg/day, once daily dose, tablets, orally
  Absolute values at Week 12 in Period 2 (Study Week 24)
Arm/Group | Period 2 Absolute Mean at Baseline; Placebo and PAR/SER | Period 2 Absolute Mean at Baseline; Brexpiprazole and PAR/SER | Period 2 Absolute Mean at Week 12; Placebo and PAR/SER | Period 2 Absolute Mean at Week 12; Brexpiprazole and PAR/SER
Number analyzed (Participants) | 17 | 23 | 15 | 17
Score | 82.82 (12.94) | 83.43 (13.12) | 69.67 (20.26) | 69.18 (18.17)

2. Secondary Outcome: Global Clinical Impression Severity of Illness (CGI-S) Score
Description: Clinical Global Impression - Severity of Illness (CGI-S) The CGI-S provides the clinician's impression of the patient's current state of mental illness. The clinician uses his or her clinical experience of this patient population to rate the severity of the patient's current mental illness on a 7-point scale ranging from 1 (Normal - not at all ill) to 7 (among the most extremely ill patients).
Time Frame: Period 2: Baseline to Week 12 (of randomized period)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score
Groups:
- Period 2 Absolute Mean at Week 12; Placebo and PAR/SER: Period 2 absolute mean value at Week 12; Randomized placebo adjunct to open-label treatment with a commercially available approved treatment for PTSD (PAR/SER) Placebo: Once daily, tablets, orally Absolute values at Week 12 in Period 2 (Study Week 24); randomized period.
- Period 2 Absolute Mean at Week 12; Brexpiprazole and PAR/SER: Period 2 absolute mean value at Week 12; Randomized brexpiprazole adjunct to open-label treatment with a commercially available approved treatment for PTSD (PAR/SER); randomized period.
  Brexpiprazole dosing was 1mg/day for one week, followed by 2mg/day for 3 weeks. Thereafter the dose was flexible and could be adjusted from 1 to 3 mg/day. Brexpiprazole: 1 to 3 mg/day, once daily dose, tablets, orally Absolute values at Week 12 in Period 2 (Study Week 24).
Arm/Group | Period 2 Absolute Mean at Baseline; Placebo and PAR/SER | Period 2 Absolute Mean at Baseline; Brexpiprazole and PAR/SER | Period 2 Absolute Mean at Week 12; Placebo and PAR/SER | Period 2 Absolute Mean at Week 12; Brexpiprazole and PAR/SER
Number analyzed (Participants) | 17 | 23 | 15 | 17
Score | 4.24 (0.83) | 4.54 (0.73) | 3.73 (1.10) | 3.94 (0.83)

ADVERSE EVENTS:
Time Frame: Period 2: Baseline to Week 16 (randomized period)
Arm/Group | Brexpiprazole + PAR/SER (Randomized Period) | Placebo + PAR/SER (Randomized Period)
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/17
Other Adverse Events (participants affected / at risk) | 3/23 | 8/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole + PAR/SER (Randomized Period) (N=23) | Placebo + PAR/SER (Randomized Period) (N=17)
Conjunctivitis (Eye disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 2 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Disturbance in attention (Nervous system disorders) | 0 | 1
Galactorrhoea (Reproductive system and breast disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
As the study was terminated limited efficacy and safety data were collected from the randomized patients. The data are descriptive and the primary and key secondary efficacy analyses were not done.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No